CLINICAL TRIAL: NCT06087978
Title: A Phase 1, Open-Label Study to Characterize the Absorption, Metabolism, Excretion (ADME), and Mass Balance of a Single Oral Dose of [14C]-RPT193 in Healthy Adult Male Subjects
Brief Title: Study of RPT193 in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RAPT Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RPT193-04
Record Dates: First submitted 2023-10-04; First posted 2023-10-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 14C RPT193 400 mg (Experimental): Radiolabelled RPT193
  Interventions: Drug: 14C RPT193

INTERVENTIONS:
Drug: 14C RPT193 — Radiolabelled RPT193

SUMMARY:
Phase 1, open-label, absorption, metabolism, excretion, and mass balance study.

DETAILED DESCRIPTION:
A study of RPT193 in healthy volunteers to evaluate the route(s) of elimination and overall mass balance of RPT193 in urine and feces

ELIGIBILITY:
Inclusion Criteria:

* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to dosing
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at the screening

Exclusion Criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit
* History or presence of clinically significant medical or psychiatric condition or disease
* History or presence of alcohol or drug abuse within the past 2 years prior to dosing
* History or presence of:

  * Gastrointestinal ulcers, or history of other significant GI diseases
  * Malignancy within the last 5 years, with the exception of successfully treated basal cell carcinoma.
  * Clinically significant history of angina, myocardial infarction, syncope, clinically significant cardiac arrhythmias, left ventricular hypertrophy, cardiomyopathy, or any other cardiovascular abnormality
  * Ongoing or recent (within 30 days prior to RPT193 administration) bacterial, fungal, or viral infection requiring therapy
  * Known family history of sudden death.
* Positive for human immunodeficiency virus, hepatitis B, hepatitis C
* Unwilling to abstain from alcohol, xanthane-containing beverages or food or foods containing grapefruit/Seville orange prior to admission
* Received radiolabeled substances or exposed to radiation sources over past 12 months

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Route(s) of elimination 1 | 14 days
  Amount (in mass equivalents of parent drug) of radioactive drug excreted as TRA in urine and feces
Route(s) of elimination 2 | 14 days
  Percent (%) of radioactive drug excreted as TRA in urine and feces
Quantitate total radioactivity (TRA) | 14 days
  Percent (%) of each drug-related material (parent and each metabolite) in whole blood, plasma, urine and feces
Characterize pharmacokinetics (PK) profile of RPT193 | 14 days
  Calculation of area under the curve (AUC) in plasma and urine
Characterize pharmacokinetics (PK) profile of RPT193 | 14 days
  Calculation of peak plasma concentration (Cmax) in plasma and urine
Characterize pharmacokinetics (PK) profile of RPT193 | 14 days
  Calculation of time to peak plasma concentration (Tmax) in plasma and urine
Characterize pharmacokinetics (PK) profile of RPT193 | 14 days
  Calculation of half-life in plasma and urine
Characterize pharmacokinetics (PK) profile of RPT193 | 14 days
  Calculation of elimination constant in plasma and urine

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States